CLINICAL TRIAL: NCT02446392
Title: The Distribution of Plasma Drug Concentrations of Beta-lactam Antibiotics in Intensive Care Unit Patients
Acronym: TDM-ICU
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Thomas Schon, MD PhD (Associate professor), Linkoeping University
Other Study IDs: TDM-ICU
Record Dates: First submitted 2015-04-24; First posted 2015-05-18 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples at three consecutive days for measurement of plasma drug concentrations
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention.

SUMMARY:
In this project, intensive care unit (ICU) patients treated with beta-lactam antibiotics are included with the aim to investigate the potential underdosing in this patient group. Four regional ICU-clinics are recruiting consecutive patients (n=120) and samples are taken before the next dose is administered for three consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Current treatment with beta-lactam antibiotics and admission to the ICU

Exclusion Criteria:

* Pregnancy, age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care unit patients treated with beta-lactam antibiotics
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The rate of patients below 16mg/L for piperacillin-tazobactam, 2 mg/L for meropenem and 4mg/L for cefotaxim | 3 days

SECONDARY OUTCOMES:
Mortality in relation to initial levels of beta-lactam antibiotics as defined in primary outcome | 30 days
The rate of patients below 100% time over MIC in relation to the bacteria causing the infection. | 3 days
Kidney function measured as eGFR in relation to initial levels of beta-lactam antibiotics as defined in primary outcome | 3 days
SAPS-score in relation to initial levels of beta-lactam antibiotics as defined in primary outcome | 3 days
Days in intensive care unit in relation to initial levels of beta-lactam antibiotics as defined in primary outcome | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schön, MD PhD, Principal Investigator — Linkoeping University
Locations (4):
- Sweden (4):
  - Intensive care unit, Jönköping, Jönköping County
  - Intensive Care Unit, Kalmar, Kalmar County
  - Intensive Care Unit, Linköping, Linköping
  - Intensive care unit, Vaxjo, Växjö

REFERENCES:
- [Background] Udy AA, Roberts JA, Lipman J. Clinical implications of antibiotic pharmacokinetic principles in the critically ill. Intensive Care Med. 2013 Dec;39(12):2070-82. doi: 10.1007/s00134-013-3088-4. Epub 2013 Sep 18. PMID 24045886